CLINICAL TRIAL: NCT01356472
Title: Linezolid Alone or Combined With Carbapenem Against Methicillin-resistant Staphylococcus Aureus (MRSA) in Vitro and in Ventilator-associated Pneumonia
Brief Title: Linezolid Alone or Combined With Carbapenem Against Methicillin-resistant Staphylococcus Aureus (MRSA) in Ventilator-associated Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: YANG Zhi-Tao, Emergency Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRSA-VAP YANG ZT CN
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-04

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Pneumonia, Ventilator-Associated
Keywords: Methicillin-resistant Staphylococcus aureus; Pneumonia, Ventilator-Associated; linezolid; imipenem/cilastatin
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Linezolid alone (No Intervention): the control group is designed for linezolid alone treated MRSA VAP (standard treatment).
  Interventions: Drug: Imipenem/cilastatin

INTERVENTIONS:
Drug: Imipenem/cilastatin — the intervention group was designed for combined linezolid plus imipenem for treating MRSA VAP

SUMMARY:
As previous studies showed that the synergy between linezolid and carbapenem in vitro and in vivo (animal studies), our study is aim to investigate the activity of linezolid, alone and in combination with carbapenem against methicillin-resistant Staphylococcus aureus (MRSA) in ventilator-associated pneumonia (VAP) patients.

DETAILED DESCRIPTION:
Linezolid is the only commercially available oxazolidinone, the first new class of antibiotic to be developed in the last three decades. Although it is predominantly bacteriostatic, linezolid has good in vitro and in vivo activity against MRSA . However, several studies did not show that linezolid was superior to any of glycopeptides in treatment of MRSA pneumonia. Moreover, combination therapy against MRSA is argued when several in vitro and in vivo studies showed synergy between linezolid and carbapenem or fosfomycin or rifampicin, while vancomycin and linezolid in combination should be avoided. our study is aim to investigate the activity of linezolid, alone and in combination with carbapenem against methicillin-resistant Staphylococcus aureus (MRSA) in ventilator-associated pneumonia (VAP) patients.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia, Ventilator-associated

  * the presence of new or persistent radiographic features
  * fever higher than 38°C
  * leukocytosis (≥11.0 ×109/L) or neutropenia (≤3.5×109/L)
  * purulent endotracheal
  * increasing oxygen requirements
* Endotracheal aspiration culture show methicillin-resistant S. aureus positive

Exclusion Criteria:

* immunocompromised patients (postorgan transplantation or human immunodeficiency virus-infected or neutropenic [≤1×109/L absolute neutrophils], or patients receiving corticosteroids >20 mg/d for 6 months)
* colonized chronically with methicillin-resistant S. aureus
* pregnancy
* endotracheal aspiration culture showed no MRSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
MRSA eradication | 7 th day
  The investigators study the efficacy of Linezolid combined with Imipenem to treat the MRSA VAP, the investigators proposed the 7th day's MRSA eradication would be better than Linezolid alone.

SECONDARY OUTCOMES:
MRSA eradication | 14th day
mortality | 28th day

CONTACTS AND LOCATIONS:
Overall Officials: Er-Zhen Chen, M.D. & Ph.D., Study Director — Emergency intensive care unit, Ruijin Hospital; Hong-Ping Qu, M.D., Principal Investigator — Respiratory intensive care unit, Ruijin Hospital; Yu-Xing Ni, M.D. & Ph.D., Principal Investigator — Microbiology laboratory, Ruijin Hospital; Zhi-Tao Yang, M.D., Study Chair — Emergency Department, Ruijin Hospital

REFERENCES:
- [Background] Jacqueline C, Navas D, Batard E, Miegeville AF, Le Mabecque V, Kergueris MF, Bugnon D, Potel G, Caillon J. In vitro and in vivo synergistic activities of linezolid combined with subinhibitory concentrations of imipenem against methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 2005 Jan;49(1):45-51. doi: 10.1128/AAC.49.1.45-51.2005. PMID 15616274
- [Background] Jacqueline C, Caillon J, Grossi O, Le Mabecque V, Miegeville AF, Bugnon D, Batard E, Potel G. In vitro and in vivo assessment of linezolid combined with ertapenem: a highly synergistic combination against methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 2006 Jul;50(7):2547-9. doi: 10.1128/AAC.01501-05. PMID 16801442
- [Background] Rubinstein E, Cammarata S, Oliphant T, Wunderink R; Linezolid Nosocomial Pneumonia Study Group. Linezolid (PNU-100766) versus vancomycin in the treatment of hospitalized patients with nosocomial pneumonia: a randomized, double-blind, multicenter study. Clin Infect Dis. 2001 Feb 1;32(3):402-12. doi: 10.1086/318486. Epub 2001 Jan 26. PMID 11170948
- [Background] Shorr AF, Kunkel MJ, Kollef M. Linezolid versus vancomycin for Staphylococcus aureus bacteraemia: pooled analysis of randomized studies. J Antimicrob Chemother. 2005 Nov;56(5):923-9. doi: 10.1093/jac/dki355. Epub 2005 Sep 29. PMID 16195255
- [Background] Stevens DL, Herr D, Lampiris H, Hunt JL, Batts DH, Hafkin B. Linezolid versus vancomycin for the treatment of methicillin-resistant Staphylococcus aureus infections. Clin Infect Dis. 2002 Jun 1;34(11):1481-90. doi: 10.1086/340353. Epub 2002 May 13. PMID 12015695